CLINICAL TRIAL: NCT06505863
Title: Does Transanal Total Mesorectal Excision (taTME) Result in Better Quality of Life and Functional Outcomes Than Traditional Total Mesorectal Excision? A Retrospective Propensity Score-adjusted Cohort Study
Brief Title: Quality of Life After Transanal Total Mesorectal Excision Compared to Traditional Total Mesorectal Excision
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Yanic Ammann, Dr. med., Cantonal Hospital of St. Gallen
Other Study IDs: taTME QoL
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Quality of Life; Functional Outcome; Surgery
Keywords: Transanal total mesorectal excision; Laparoscopic total mesorectal excision
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- taTME: Patients who underwent transanal total mesorectal excision with anastomosis for primary rectal cancer UICC stage I to III
  Interventions: Procedure: Transanal total mesorectal excision
- abTME: Patients who underwent laparoscopic, robotic, or open total mesorectal excision with anastomosis for primary rectal cancer UICC stage I to III
  Interventions: Procedure: Abdominal total mesorectal excision

INTERVENTIONS:
Procedure: Transanal total mesorectal excision — Transanal approach in surgical treatment of rectal cancer along the anatomical and embryological planes, called total mesorectal excision, as described in 1988 by Heald et al.
  Groups: taTME
Procedure: Abdominal total mesorectal excision — Patients who underwent laparoscopic, robotic, or open total mesorectal excision with anastomosis for primary rectal cancer UICC stage I to III
  Groups: abTME

SUMMARY:
The improvement in prognosis of rectal cancer through modern therapy modalities rises questions regarding quality of life (QoL) and functional outcomes. Evidence for long-term QoL and functional outcomes of transanal total mesorectal excision (taTME) is not provided in current literature. This study will compare short-term and long-term QoL and functional outcomes after taTME compared to traditional abdominal TME (laparoscopic, robotic, and open approach)

DETAILED DESCRIPTION:
Quality of life and functional outcomes of patients undergoing taTME or abTME for stage I-III rectal cancer will be analysed. A retrospective propensity score-adjusted analysis of prospectively conducted data will be performed. The primary endpoint QoL will be assessed by the European Organization for Research and Treatment of Cancer core questionnaire (EORTC QLQ-C30). Secondary endpoints are the functional outcomes according to the EORTC QLQ-C30 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* elective total mesorectal excision followed by reconstruction with anastomosis for primary rectal cancer

Exclusion Criteria:

* diagnoses other than rectal cancer
* recurrent rectal cancer
* partial mesorectal excision
* discontinuity resection (no anastomosis)
* incomplete TNM staging information
* metastatic cancer
* 30-day mortality
* lack of quality of life data
* patient decline
* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving elective total mesorectal excision followed by reconstruction with anastomosis for primary rectal cancer at the Cantonal hospital of St.Gallen, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) | 5 years after initial operation
  Assessed by the European Organization for Research and Treatment of Cancer core questionnaire (EORTC QLQ-C30):
  * Overall QoL
  * QLQ-total

SECONDARY OUTCOMES:
Functional outcomes | 5 years after initial operation
  Assessed by the European Organization for Research and Treatment of Cancer core questionnaire (EORTC QLQ-C30):
  * physical functioning
  * role functioning
  * cognitive functioning
  * emotional functioning
  * social functioning
  * fatigue
  * pain
  * nausea and vomiting
  * appetite loss
  * dyspnea
  * insomnia
  * constipation
  * diarrhea
  * financial difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Walter Brunner, PD Dr. med., Study Director — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital of St.Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No
The anonymized patient data that support the findings of this study are available and can be obtained upon reasonable request.

REFERENCES:
- [Background] Heald RJ. The 'Holy Plane' of rectal surgery. J R Soc Med. 1988 Sep;81(9):503-8. doi: 10.1177/014107688808100904. No abstract available. PMID 3184105
- [Derived] Ammann Y, Klein M, Marti L, Warschkow R, Strose L, Sparn M, Jager T, Bischofberger S, Brunner W. Does transanal total mesorectal excision (taTME) result in better quality of life and functional outcomes than traditional TME does? A retrospective propensity score-adjusted cohort study. Langenbecks Arch Surg. 2025 Apr 30;410(1):149. doi: 10.1007/s00423-025-03724-6. PMID 40304801